CLINICAL TRIAL: NCT03281551
Title: Study of Anti-CD19 Chimeric Antigen Receptor T Cells（PZ01） for Relapsed/ Refractory B-cell Acute Lymphoblastic Leukemia/B Cell Lymphoma
Brief Title: Efficacy and Safety of PZ01 Treatment in Patients With r/r CD19+ B-cell Acute Lymphoblastic Leukemia/B Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pinze Lifetechnology Co. Ltd. (Industry)
Collaborators: Chinese Academy of Sciences (Other Government); Navy General Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PZ01
Record Dates: First submitted 2017-09-09; First posted 2017-09-13 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: B-cell Acute Lymphoblastic Leukemia; B-cell Lymphoma
MeSH Terms: conditions — Burkitt Lymphoma; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PZ01 CAR-T Cells (Experimental): This is a phase I study. Patients with relapsed/ refractory B-cell Acute Lymphoblastic Leukemia/B cell Lymphoma are eligible for enrollment.
  Interventions: Drug: PZ01 CAR-T cells

INTERVENTIONS:
Drug: PZ01 CAR-T cells — Chimeric antigen receptor (CAR) T cells targeting CD19 will be evaluated for safety and efficacy in patients with relapsed/ refractory B-cell Acute Lymphoblastic Leukemia/B cell Lymphoma. The CAR consists of a CD19 targeting antibody scFv with two intracellular signaling domains derived from CD3 zeta and 4-1BB. Autologous T cells will be gene-engineered with the CAR gene using a lentivirus vector. Prior to T cell infusion, the patients will be subjected to preconditioning treatment. After T cell infusion, the patients will be evaluated for 24 months for adverse reactions, persistence of CAR T cells and efficacy.

SUMMARY:
The major aim of this research is to assess the feasibility, safety and effectiveness of CD19 CAR-T Cell Therapy for Relapsed/ Refractory Acute Lymphoblastic Leukemia/ B cell Lymphoma patients who have applied it.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects or their legal guardians participate in this experiment voluntarily and informed consent form must be signed
2. In accordance with National Comprehensive Cancer Network (NCCN) ALL Guidelines for Patients (2016, v.1) and CD19+B-ALL/B cell lymphoma patients diagnosed by histology
3. In accordance with r/r CD19+ B-ALL/B cell lymphoma diagnosis, including any of the following situations:

   1. Getting through 2 treatments of standard chemotherapy with CR not yet obtained
   2. Reach CR for the first inducement, but CR lasts for ≦12 months
   3. r/r CD19+ B-ALL/B cell lymphoma for no positive effect after first or repeated remedial treatment
   4. ≧2 times of recurrence
4. Remedial chemotherapy is not used within 4 weeks before cell therapy
5. Immunosuppressive drug is not used within 4 weeks before cell therapy, including but not limited to systemic hormone therapy
6. Antibody drug treatment is not received within 2 weeks before cell therapy
7. Normal cardiac motion shown by echocardiography, left ventricular ejection fraction (LVEF) ≥50%, with no pericardial effusion and severe symptoms of cardiac arrhythmia
8. No pulmonary active infection is found, with normal pulmonary function and indoor air SaO2 ≧92%
9. No contraindications for leukapheresis
10. Expected survival >3 months
11. Grade 0 or 1 of ECOG performance status

Exclusion Criteria:

1. Pregnant and breastfeeding women
2. Uncontrolled active infection
3. Uncontrolled infectious disease is diagnosed, such as HIV, syphilis, hepatitis A, hepatitis B, hepatitis C and E.
4. Patients who have used a large amount of glucocorticoid or other immunosuppressive drugs within 4 weeks
5. Stage II-IV Acute/chronic general graft versus host disease
6. Gene therapy has been undergone in the past

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related Adverse Events | 1 year
  To evaluate the safety of adoptive transfer of gene-modified autologous CD19-specific T cells in relapsed/ refractory B-cell Acute Lymphoblastic Leukemia/B cell Lymphoma.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 months
  Proportion of patients with reduction in tumor burden.
Overall survival (OS) | 6 months
  Time from study enrollment until death.
Minimal residual disease negative remission rate(MRD) | 2 months
  Proportion of MRD-negative patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shengdian Wang, Principal Investigator — Insitute of Biophysics,Chinese Academy of Sciences
Locations (1):
- Department of Hematology, Navy General Hospital of PLA, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No